CLINICAL TRIAL: NCT01078974
Title: Phase I Study of Pomalidomide, Dexamethasone and Rituximab (PDR) in Relapsed or Refractory Waldenstrom's Macroglobulinemia
Brief Title: Pomalidomide, Dexamethasone and Rituximab in Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety concerns (IgM Flare)
Sponsor: Steven P. Treon, MD, PhD (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Steven P. Treon, MD, PhD, Principal Investigator, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-007; PO-WM-PI-0005 (Other: Celgene)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: WM; pomalidomide; dexamethasone; rituximab
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — pomalidomide; Dexamethasone; Calcium Dobesilate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pomalidomide, dexamethasone, rituximab (Experimental): Drug: pomalidomide Taken orally once a day
  Drug: dexamethasone Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
  Drug: rituximab Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
  Interventions: Drug: pomalidomide; Drug: dexamethasone; Drug: rituximab

INTERVENTIONS:
Drug: pomalidomide — Taken orally once a day
  Other Names: CC-4047; Pomalyst
Drug: dexamethasone — Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
  Other Names: Decadron
Drug: rituximab — Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
  Other Names: Rituxan

SUMMARY:
Pomalidomide is a newly discovered drug that may stop cancer cells from growing abnormally. Pomalidomide may also stimulate the immune system to fight the cancer cells and possibly improve the effectiveness of dexamethasone and rituximab to fight the Waldenstrom's Macroglobulinemia (WM) cancer cells. This drug have been used in multiple myeloma and information from these other research studies suggests that Pomalidomide may help to reduce or prevent the growth of cancer cells.

DETAILED DESCRIPTION:
* Participants will be given a study drug-dosing calendar for each treatment cycle. Each treatment cycle lasts 28 days during which time participants will take Pomalidomide orally once a day. Dexamethasone and rituximab will be administered intravenously on weeks 1, 2, 3, 4 and on weeks 12, 13, 14, 15.
* Since we are looking for the highest dose of Pomalidomide in combination with dexamethasone and rituximab which can be administered safely without severe or unmanageable side effects, not everyone who participates will receive the same dose of the study drug. The dose participants will get will depend on the number of participants who have been enrolled in the study and how well they have tolerated their doses.
* As long as there is no evidence that the participant's Waldenstrom's Macroglobulinemia has progressed, they can continue to receive Pomalidomide for up to 52 weeks. Participants will be asked to return to the clinic for follow-up tests at least every three months for four years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to adhere to the study visit schedule and other protocol requirements
* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia using consensus panel criteria
* CD20 positive based on any previous performed bone marrow immunohistochemistry or flow cytometric analysis
* Meet criteria to treat based on consensus panel criteria
* Patient must have received at least one previous therapy for WM
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level of 2 times (or greater) the upper limit of each institution's normal value is required
* ECOG Performance status of 0, 1 or 2
* Laboratory tests within ranges outlined in the protocol
* Disease free of prior malignancies for 5 years or more with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast
* Screening of patients at high risk of HBV or HCV infection
* Willing and able to take aspirin or alternate prophylactic anticoagulants

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness
* Pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Resistance or intolerance to prior rituximab therapy
* Previous therapy with thalidomide or lenalidomide
* Known hypersensitivity to thalidomide, lenalidomide or pomalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking similar drugs
* Concurrent use of other anti-cancer agents or treatments
* History of non-compliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Known positive for HIV or hepatitis infection
* Any history of CVA (Cerebral Vascular Accident/stroke) or clots
* Active DVT or PE that has not been therapeutically anticoagulated
* NYHA classification III and greater heart failure
* Any patient that is unable to ingest or process pomalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-05; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Treon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 7 participants were recruited at the DFCI medical clinic between 9/22/2010 and 4/3/2012.
Groups:
- Pomalidomide, Dexamethasone, Rituximab: Drug: pomalidomide Taken orally once a day
  Drug: dexamethasone Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
  Drug: rituximab Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
  pomalidomide: Taken orally once a day
  dexamethasone: Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
  rituximab: Given intravenously on weeks 1, 2, 3 and 4 and weeks 12, 13, 14 and 15
Period: Overall Study
Arm/Group | Pomalidomide, Dexamethasone, Rituximab
Started | 7
Completed | 4
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pomalidomide, Dexamethasone, Rituximab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Median (Standard Deviation); unit: years] | 64 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Pomalidomide
Description: To determine the MTD of pomalidomide administered orally in patients with Waldenstrom's Macroglobulinemia in combination with dexamethasone and rituximab. Because maximum tolerated dose was not determined due to study termination, the highest dose of pomalidomide administered is presented below.
Time Frame: 2 years
Population: The maximum tolerated dose was not determined due to study termination. Three participants experienced IgM flare causing them to be removed from the study early.
Measure: Number; unit: mg
Arm/Group | Pomalidomide, Dexamethasone, Rituximab
Number analyzed (Participants) | 7
mg | 1

2. Primary Outcome: Tolerability of Pomalidomide
Description: Number of participants with dose limiting toxicities which resulted in being removed from pomalidomide therapy
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Pomalidomide, Dexamethasone, Rituximab
Number analyzed (Participants) | 7
participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 3 year period.
Arm/Group | Pomalidomide, Dexamethasone, Rituximab
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide, Dexamethasone, Rituximab (N=7)
IgM flare (Blood and lymphatic system disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide, Dexamethasone, Rituximab (N=7)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Cough (General disorders) | 1 (1)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
INR increased (Metabolism and nutrition disorders) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (3)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (3)
Seizure (Nervous system disorders) | 1 (2)
Tooth Infection (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Urinary frequency (General disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Pomalidomide and rituximab could have a synergistic effect on serum IgM levels and produce an IgM flare. The highest dose of pomalidomide in this trial was 1mg. The study was permanently closed to accrual given the safety concerns with the IgM flare.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes